CLINICAL TRIAL: NCT04727645
Title: Prospective Use of Philips "iSuite" Electroanatomical Mapping System in Addition to Standard CMR-guided Electrophysiological Procedures
Brief Title: Use of "iSuite" During CMR-guided Electrophysiological Procedures
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Academisch Ziekenhuis Maastricht (Other)
Responsible Party: Principal Investigator, S.M. Chaldoupi, MD, PhD, Academisch Ziekenhuis Maastricht
Other Study IDs: NL74812.068.20; METC20-064 (Other: METC azM/UM)
Record Dates: First submitted 2021-01-18; First posted 2021-01-27 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-02

CONDITIONS: Cardiac Arrhythmia
Keywords: Cardiac Magnetic Resonance Imaging (CMR); CMR-guided electrophysiological procedure; Radiofrequency ablation
MeSH Terms: conditions — Arrhythmias, Cardiac | interventions — Bestrophins

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Philips interventional MRI suite (Philips Healthcare, Best, the Netherlands) — iSuite is an an electroanatomical mapping system (EAM) designed to support real-time MRI guided interventional procedures.
  Other Names: "iSuite"

SUMMARY:
The perpuse of this study is to investigate the feasibility of the Philips interventional MRI suite "iSuite" to create an electroanatomical map of the heart based on which the real-time location of the catheters can be correctly and reliably visualized during CMR-guided electrophysiological procedure (CMR-EP).

ELIGIBILITY:
Inclusion Criteria:

* Already scheduled by the treating electrophysiologist for CMR-EP as standard care for the treatment of a cardiac arrhythmia.
* Minimum age of 18 years old.
* Written informed consent

Exclusion Criteria:

* Participation in another investigational study that has not reached its primary endpoint.
* Contraindication for MRI such as: metallic implant, body weight > 130 kg, pregnancy, breast feeding women, known severe allergy to gadolineum contrast agents, renal failure with eGFR ≤ 30 mL/min/1,73m2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include all eligible patients who are already scheduled and thus eligible for CMR-guided electrophysiological procedure for the treatment of a cardiac rhythm disturbance in the MUMC+, albeit meeting the in- and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-01-04 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
The feasibility of iSuite to create an electroanatomical map (EAM) of the heart during CMR-EP | Periprocedural
  To establish whether the visualization by iSuite is correct we will compare the location visualized by the EAM with the reference images as produced by the default cine MRI sequences at the target ablation location just prior to the RF ablation. The definition of correct visualization is: good agreement between the two modalities (EAM and cine MRI) based on visual assessment of the treating electrophysiologist and the supervising CMR expert. When no consensus is reached than the visualization is coded 'incorrect'. This outcome will be dichotomized and coded as 'correct visualization' or 'incorrect visualization'. This categorical variable will be expressed as counts and proportion with 95% confidence interval (CI).

SECONDARY OUTCOMES:
Procedural success as measured by electrical and anatomical confirmation of a complete ablation lesion at the end of the procedure: | Periprocedural
  Anatomical confirmation of a complete ablation lesion is defined as a continuous line of high signal intensity at the target location on the edema and fibrosis sequences of the CMR at the end of the procedure. This anatomical confirmation will be judged by the CMR expert that is present during the procedure and thus will not be blinded to the EP results. Procedural success and procedural complications will be reported as count and proportion with 95% CI.
Procedural time | Periprocedural
  To investigate the procedure-by-procedure change in procedural times and total amount of CMR images needed until application of the first ablation lesion
Complication rate | Periprocedural
  To investigate the complication rate of CMR-EP with the integration of iSuite.

CONTACTS AND LOCATIONS:
Overall Officials: S.M. Chaldoupi, Principal Investigator — Maastricht UMC; Casper Mihl, Principal Investigator — Maastricht UMC; J.E Wildberger, Prof. Dr, Study Chair — Maastricht UMC
Locations (1):
- Maastricht UMC+, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No
This is a small scale single center study and there is no plan to share IPD in order to ensure participant privacy, and the risk of invalid analysis. Data will be registered in the Castor EDC database by the investigator, after patient data has been anonymized. The principal investigator and involved investigators of the research team will have access to the source data and safeguard the code. The handling of personal data will comply with the General Data Protection Regulation and the Dutch Act on Implementation of the General Protection Regulation. Data and the key to the unique patient study number will be kept for 15 years after study end. During this single centre study, no data will be shared or transferred. Once the study has ended, we will ensure that all data are managed and securely stored. Data will be available for use in future research on cardiac arrhythmia. Qualified monitors of Clinical Trial Centre Maastricht will independently perform monitoring of the study.

REFERENCES:
- [Background] Hilbert S, Sommer P, Gutberlet M, Gaspar T, Foldyna B, Piorkowski C, Weiss S, Lloyd T, Schnackenburg B, Krueger S, Fleiter C, Paetsch I, Jahnke C, Hindricks G, Grothoff M. Real-time magnetic resonance-guided ablation of typical right atrial flutter using a combination of active catheter tracking and passive catheter visualization in man: initial results from a consecutive patient series. Europace. 2016 Apr;18(4):572-7. doi: 10.1093/europace/euv249. Epub 2015 Aug 27. PMID 26316146
- [Background] Paetsch I, Sommer P, Jahnke C, Hilbert S, Loebe S, Schoene K, Oebel S, Krueger S, Weiss S, Smink J, Lloyd T, Hindricks G. Clinical workflow and applicability of electrophysiological cardiovascular magnetic resonance-guided radiofrequency ablation of isthmus-dependent atrial flutter. Eur Heart J Cardiovasc Imaging. 2019 Feb 1;20(2):147-156. doi: 10.1093/ehjci/jey143. PMID 30307544
- [Background] Vergara GR, Vijayakumar S, Kholmovski EG, Blauer JJ, Guttman MA, Gloschat C, Payne G, Vij K, Akoum NW, Daccarett M, McGann CJ, Macleod RS, Marrouche NF. Real-time magnetic resonance imaging-guided radiofrequency atrial ablation and visualization of lesion formation at 3 Tesla. Heart Rhythm. 2011 Feb;8(2):295-303. doi: 10.1016/j.hrthm.2010.10.032. Epub 2010 Oct 27. PMID 21034854
- [Background] Lichter J, Kholmovski EG, Coulombe N, Ghafoori E, Kamali R, MacLeod R, Ranjan R. Real-time magnetic resonance imaging-guided cryoablation of the pulmonary veins with acute freeze-zone and chronic lesion assessment. Europace. 2019 Jan 1;21(1):154-162. doi: 10.1093/europace/euy089. PMID 29878090